CLINICAL TRIAL: NCT02723682
Title: National Health and Nutrition Examination Survey 24-Hour Urine Collection Feasibility Study, 2013
Status: Completed | Type: Observational
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2011-17
Record Dates: First submitted 2016-03-08; First posted 2016-03-30 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Collect 24-hour urine specimen — A random half sample of NHANES participants 20-69 examined in the mobile examination center were asked to collect a 24-hour urine specimen.

SUMMARY:
A 24-hour urine pilot study was conducted as part of the 2013 NHANES to test the feasibility of implementing a 24-hour urine collection as part of NHANES in 2014.

DETAILED DESCRIPTION:
The 24-hour urine pilot study was conducted March - June 2013 in three NHANES locations. A random half-sample of non-pregnant US adults, aged 20-69 who were examined in the NHANES mobile examination center were selected. Participants received instructions, started and ended the urine collection in a urine study mobile examination center (UMEC), and answered questions about collection. A random half of participants who collected a complete 24-h urine were asked to collect a second 24-h urine. Urinary sodium, potassium, chloride, and creatinine excretion were analyzed.

Participation rates in two other post-examination components, the Physical Activity Monitor and the Dietary Recall, were monitored to determine whether collecting a 24-hour urine had an effect on response rates for the two components.

ELIGIBILITY:
Inclusion Criteria:

* 20-69 year old adults examined in the NHANES mobile examination center

Exclusion Criteria:

* pregnant, unable to respond for themselves

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: NHANES participants aged 20-69 years who were examined in the mobile examination center.
Sampling Method: Probability Sample
Enrollment: 282 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Study completion rates - initial collection | 24 hours
  Completion rate of initial 24-hour urine collection.
Study completion rate - second collection | 24 hours
  Completion rate of second 24-hour urine collection

SECONDARY OUTCOMES:
Response rates for the Physical Activity Monitor | 24-hours
  Response rates for the Physical Activity Monitor
Response rates for the Phone Follow-up Dietary Recall | 24-hours
  Response rates for the Phone Follow-up Dietary Recall.
Urine volume for the initial urine collection | 24 hours
  Urine volume adjusted to 24 hours, initial urine collection
Urine volume for the second urine collection | 24 hours
  Urine volume adjusted to 24 hours, second urine collection
Urinary sodium excretion for the initial urine collection | 24 hours
  24-hour urinary sodium excretion, initial urine collection
Urinary sodium excretion for the second urine collection | 24 hours
  24-hour urinary sodium excretion, second urine collection

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Porter, MD, MS, Study Director — Centers for Disease Control and Prevention, National Center for Health Statistics, Division of Health and Nutrition Examination Surveys
Locations (1):
- National Health and Nutrition Examination Survey, Hyattsville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
The NHANES 24-hour urine pilot study data set can be made available through the National Center for Health Statistics Research Data Center by submitting a research proposal at http://www.cdc.gov/rdc/.

REFERENCES:
- [Derived] Terry AL, Cogswell ME, Wang CY, Chen TC, Loria CM, Wright JD, Zhang X, Lacher DA, Merritt RK, Bowman BA. Feasibility of collecting 24-h urine to monitor sodium intake in the National Health and Nutrition Examination Survey. Am J Clin Nutr. 2016 Aug;104(2):480-8. doi: 10.3945/ajcn.115.121954. Epub 2016 Jul 13. PMID 27413136